CLINICAL TRIAL: NCT07323537
Title: Youtube as Sources of Information on One of the Biggest Causes of Preoperative Anxiety "Anesthesia Awareness": Assessment and Analysis of the Content and Quality.
Brief Title: Anesthesia Awareness on YouTube: Content and Quality Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: Mentese State Hospital (Other Government)
Responsible Party: Principal Investigator, Pelin Dilsiz Eker, Medical Doctor, Specialist, Mentese State Hospital
Other Study IDs: 2025-discern
Record Dates: First submitted 2025-11-19; First posted 2026-01-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Awareness, Anesthesia
Keywords: YouTube; DISCERN score; Usefullness score; Global quality score (GQS); Journal of the american medical association (JAMA) score; Patient Education Materials Assessment Tool for Audiovisual Content (PEMAT-A/V)
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the quality and reliability of YouTube videos related to "anesthesia awareness." Using the search terms "anesthesia awareness" and "waking up during surgery," the first 100 videos from each search query will be identified and their URLs recorded. After applying predefined inclusion and exclusion criteria, an eligible video list will be created for independent reviewers. Each video will be assessed using five validated scoring instruments: the modified DISCERN score, the Global Quality Scale (GQS), the JAMA benchmark criteria, the Patient Education Materials Assessment Tool for Audiovisual Content (PEMAT-A/V), and a usefulness score. The study seeks to characterize the educational value and accuracy of publicly available online content on anesthesia awareness.

ELIGIBILITY:
Inclusion Criteria:

* Videos in English language.
* Videos addressing "anesthesia awareness" or "waking up during surgery."
* Publicly available on YouTube at the time of the search.
* Within the first 100 results for each keyword search.
* Containing audio and/or visual content suitable for evaluation using the predefined scoring tools.

Exclusion Criteria:

* Non-English language videos.
* Duplicate videos.
* Videos not relevant to the topic.
* Videos shorter than 60 seconds or longer than 60 minutes.
* Videos with audio or visual issues preventing content evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Publicly available YouTube videos on the selected keywords.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall quality score of YouTube videos on anesthesia awareness | A cross-sectional YouTube search will be conducted at study initiation, and the identified videos will be evaluated over approximately two weeks.
  The reliability and accuracy of YouTube videos on "anesthesia awareness" and "waking up during surgery" will be assessed using a validated scoring tool (modified DISCERN). In this instrument, each item is scored as 1 = Yes (criterion met) or 0 = No (criterion not met), with a total score ranging from 0 to 5. Higher scores indicate more reliable content.
Overall quality score of YouTube videos on anesthesia awareness | A cross-sectional YouTube search will be conducted at study initiation, and the identified videos will be evaluated over approximately two weeks.
  The quality of YouTube videos on "anesthesia awareness" and "waking up during surgery" will be assessed using a validated scoring tool, the Global Quality Scale (GQS). In this scale, overall quality is rated on a 5-point scale ranging from 1 (very poor quality) to 5 (excellent quality).
Overall quality score of YouTube videos on anesthesia awareness | A cross-sectional YouTube search will be conducted at study initiation, and the identified videos will be evaluated over approximately two weeks.
  The reliability, transparency, and currency of YouTube videos on "anesthesia awareness" and "waking up during surgery" will be assessed using a validated scoring tool, the Journal of the American Medical Association (JAMA) benchmark criteria. In this tool, four criteria are evaluated, with total scores ranging from 0 to 4, where 4 indicates the highest level of reliability and 0 indicates low reliability.
Overall quality score of YouTube videos on anesthesia awareness | A cross-sectional YouTube search will be conducted at study initiation, and the identified videos will be evaluated over approximately two weeks.
  The understandability and actionability of YouTube videos on "anesthesia awareness" and "waking up during surgery" will be assessed using a validated scoring tool, the Patient Education Materials Assessment Tool for Audiovisual Materials (PEMAT-A/V). In this tool, each item is scored as 1 = Agree, 0 = Disagree, or Not Applicable (N/A).
  In this instrument, score calculation is performed as follows:
  The understandability score (%) is calculated as (the total number of items scored as "1" divided by the total number of applicable items) × 100.
  The actionability score (%) is calculated as (the total number of items scored as "1" divided by the total number of applicable items) × 100.
Overall quality score of YouTube videos on anesthesia awareness | A cross-sectional YouTube search will be conducted at study initiation, and the identified videos will be evaluated over approximately two weeks.
  The educational and informational usefulness of YouTube videos on "anesthesia awareness" and "waking up during surgery" will be assessed using a validated scoring tool, the Usefulness Score. In this scale, videos are rated on a 5-point scale ranging from 1 (very low usefulness) to 5 (very high usefulness).

SECONDARY OUTCOMES:
Video View Count | Baseline
  Total number of views for each included video, will be recorded at the time of the cross-sectional YouTube search.
Video Duration | Baseline
  Length of each video in minutes and seconds.
Upload Date | Baseline
  The original upload date of each included video; used to calculate video age in days/months/years.
Engagement Metrics: Likes and Dislikes | Baseline
  Total number of likes and dislikes (if available) recorded for each video.
Comment Count | Baseline
  Number of comments posted under each included video.
Video Type Classification | Baseline
  Categorization of videos based on format: single-narrator informational video, patient experience video, animation, or slide-based presentation.
Source Classification | Baseline
  Classification of video uploaders into predefined categories: physician/hospital, non-physician healthcare personnel, medical/educational channel, or other.